CLINICAL TRIAL: NCT02556307
Title: A Study of the Effectiveness of Peginterferon Alfa-2a (Pegasys) and Ribavirin Treatment in Slovenian Hepatitis C (HCV) Patients
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22263
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Peginterferon alfa-2a + Ribavirin
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a according to the standard practice in line with current summaries \nof product characteristics (SPCs)/local labeling.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin according to the standard practice in line with current summaries \nof product characteristics (SPCs)/local labeling.
  Other Names: Copegus

SUMMARY:
In this Slovenian, multi-center, observational study, the effectiveness of standard of care Peginterferon alfa-2a + ribavirin treatment in adult patients with chronic hepatitis C (CHC) is examined. Patients were treated for 24- or 48-weeks, as prescribed by the treating physician, followed by a 24-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >/= 18 years
* Positive test for HCV
* Effective contraception as specified by the Peginterferon alfa-2a and/or ribavirin labels

Exclusion Criteria:

* Concomitant infection with HIV or hepatitis B
* Participation in a clinical trial within 30 days prior to study start
* Any contraindications specified in the Peginterferon alfa-2a and ribavirin product labels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Slovenian patients with chronic hepatitis C (CHC) treated with Peginterferon alfa-2a and ribavirin.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2009-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Slovenia (4):
  - Celje
  - Ljubljana
  - Maribor
  - Novo Mesto

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2a + Ribavirin: Participants received peginterferon alfa-2a and ribavirin according to the standard practice in line with current summaries of product characteristics (SPCs)/local labeling.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Started | 270
Treated | 268
Completed | 217
Not Completed | 53
Not completed — Premature treatment interruption | 11
Not completed — Lost to Follow-up | 36
Not completed — Change to triple therapy | 4
Not completed — Enrolled but not treated | 2

BASELINE CHARACTERISTICS:
Population: All treated participants were included in the analysis.
Groups:
- Peginterferon Alfa-2a + Ribavirin: Participants received peginterferon alfa-2a and ribavirin according to the standard practice in line with current SPCs/local labeling.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 197

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response (SVR) According to Genotype and Previous Treatment
Description: SVR was defined as participants with undetectable Hepatitis C virus (HCV) ribonucleic acid (RNA) at 24 weeks after completion of treatment. Undetectable HCV RNA was defined as a single last HCV RNA less than (<) 20 international units per milliliter (IU/mL). SVR was evaluated based on HCV genotype (G1, G2, G3 and G4), participant's interleukin 28B genotype (CC, CT and TT), and previous treatment (treatment naive or previous treatment).
Time Frame: 6 months after the last study drug administration (up to 123.6 weeks)
Population: All treated participants were included in the analysis. Here, 'n' specifies the number of participants included in the analysis as per the specified category (genotype or previous treatment).
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 268
percentage of participants
  All participants (n=268) | 66
  G1 (n=104) | 51
  G2 (n=9) | 67
  G3 (n=153) | 75
  G4 (n=2) | 100
  CC (n=56) | 66
  CT (n=73) | 66
  TT (n=25) | 64
  Treatment-naive (n=238) | 70
  Pre-treated (n=30) | 30

2. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA
Description: Undetectable HCV RNA=a single last HCV RNA <20 IU/mL
Time Frame: Weeks 4, 12 and at end of treatment (up to 99.6 weeks)
Population: All treated participants were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 268
percentage of participants
  Week 4 | 64
  Week 12 | 21
  End of treatment | 79

3. Secondary Outcome: HCV RNA Values
Time Frame: Baseline; Weeks 4, 12, end of treatment (up to 99.6 weeks) and 6 months after end of treatment (up to 123.6 weeks)
Population: Number of participants analyzed=treated participants with data available for HCV RNA. Here, "n" specifies number of participants with data available for specified category.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 267
IU/mL
  Baseline (n=267) | 3281922 (6039339)
  Week 4 (n=262) | 44174 (192056)
  Week 12 (n=219) | 21342 (189967)
  End of treatment (n=224) | 39436 (335382)
  6 months post treatment (n=195) | 93414 (852266)

4. Secondary Outcome: Thrombocyte Values
Time Frame: Baseline; Weeks 4, 12, end of treatment (up to 99.6 weeks) and 6 months after end of treatment (up to 123.6 weeks)
Population: Number of participants analyzed=treated participants with data available for thrombocyte value. Here, "n" specifies number of participants with data available for specified category.
Measure: Mean (Standard Deviation); unit: billion cells per liter
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 265
billion cells per liter
  Baseline (n=265) | 206 (62.7)
  Week 4 (n=260) | 143 (55.0)
  Week 12 (n=217) | 125 (48.0)
  End of treatment (n=224) | 140 (59.0)
  6 months post treatment (n=198) | 207 (56.0)

5. Secondary Outcome: Leukocyte Values
Time Frame: Baseline; Weeks 4, 12, end of treatment (up to 99.6 weeks) and 6 months after end of treatment (up to 123.6 weeks)
Population: Number of participants analyzed=treated participants with data available for leukocyte value. Here, "n" specifies number of participants with data available for specified category.
Measure: Mean (Standard Deviation); unit: billion cells per liter
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 265
billion cells per liter
  Baseline (n=265) | 7.0 (2.1)
  Week 4 (n=260) | 3.8 (1.4)
  Week 12 (n=217) | 3.4 (1.4)
  End of treatment (n=224) | 3.6 (1.8)
  6 months post treatment (n=198) | 7.1 (3.5)

6. Secondary Outcome: Hemoglobin Values
Time Frame: Baseline; Weeks 4, 12, end of treatment (up to 99.6 weeks) and 6 months after end of treatment (up to 123.6 weeks)
Population: Number of participants analyzed=treated participants with data available for hemoglobin. Here, "n" specifies number of participants with data available for specified category.
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 265
gram per liter
  Baseline (n=265) | 147 (14.4)
  Week 4 (n=260) | 129 (16.0)
  Week 12 (n=260) | 129 (16.0)
  End of treatment (n=224) | 122 (16.0)
  6 months post treatment (n=198) | 143 (14.0)

7. Secondary Outcome: Treatment Duration (in Weeks) With Peginterferon Alfa-2a and Ribavirin
Time Frame: Up to 99.6 Weeks
Population: All treated participants were included.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 268
weeks
  Peginterferon alfa-2a | 31.0 (17.1)
  Ribavirin | 31.3 (17.2)

ADVERSE EVENTS:
Time Frame: From signature of informed consent to end of treatment (up to 99.6 weeks)
Description: All treated participants were included.
Arm/Group | Peginterferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 4/268
Other Adverse Events (participants affected / at risk) | 15/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=268)
Headache (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Depressive disorder (Psychiatric disorders) | 1
Sudden death NOS (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=268)
Leucopenia (Blood and lymphatic system disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.